CLINICAL TRIAL: NCT00389558
Title: Comparison of Amukin Versus Biseptine Use for Dressing Application of Epicutaneocavous Catheters for Nosocomial Infection Prevention
Brief Title: Antiseptic Use and Dressing Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maternite Regionale Universitaire (Other)
Responsible Party: Prof JM HASCOET, Maternite Regionale Universitaire
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MRAP190406
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Skin Colonization; Catheterization; Bacterial Infection
Keywords: Skin colonization; Antiseptic; Epicutaneocavous catheter dressing; Infant
MeSH Terms: conditions — Bacterial Infections | interventions — Amikacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Biseptine
  Interventions: Procedure: disinfection efficacy using Biseptine
- 1 (Active Comparator): Amukin
  Interventions: Procedure: disinfection efficacy using Amukin

INTERVENTIONS:
Procedure: disinfection efficacy using Biseptine — Detersion and antiseptic application when changing catheter dressing
  Other Names: Biseptine
  Arms: 2
Procedure: disinfection efficacy using Amukin — Detersion and antiseptic application when changing catheter dressing
  Other Names: Amukin
  Arms: 1

SUMMARY:
The purposes of the study are:

1. To compare the local efficacy (skin colonization) of 2 commercialized antiseptics used for the disinfection of the dressing application for an epicutaneocavous catheter (EPI).
2. To evaluate whether the bacteria responsible for nosocomial infection is comparable to the flora diagnosed at the EPI site.

DETAILED DESCRIPTION:
Epicutaneocavous catheter is a significant risk factor for nosocomial infection in newborn infants. These infections have been related to local bacterial colonisation. Therefore thorough disinfection should lower the risk of nosocomial infection. However, the local efficacy of antiseptic use has not yet been clearly evaluated in this situation.

ELIGIBILITY:
Inclusion Criteria:

* All infants admitted to the Neonatal Intensive Care Unit
* Epicutaneocavous catheter insertion indication

Exclusion Criteria:

* Epicutaneocavous catheter not inserted within the Unit

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 453 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Efficacy on skin colonization of two commercially available antiseptics | 2 weeks

SECONDARY OUTCOMES:
In case of nosocomial infection, relationship with skin bacteria | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, Study Director — University of NANCY, France; Monique LUX, Pharmacist, Principal Investigator — Maternite Regionale Universitaire
Locations (1):
- Maternite Regionale Universitaire, Nancy, France

REFERENCES:
- [Background] Mahieu LM, De Dooy JJ, De Muynck AO, Van Melckebeke G, Ieven MM, Van Reempts PJ. Microbiology and risk factors for catheter exit-site and -hub colonization in neonatal intensive care unit patients. Infect Control Hosp Epidemiol. 2001 Jun;22(6):357-62. doi: 10.1086/501913. PMID 11519913